CLINICAL TRIAL: NCT07116031
Title: An Open-label, Phase 1/2, Multicenter Study of Belumosudil in Children Aged 1 to <18 Years Requiring Systemic Treatment for Active Moderate-to-severe Chronic Graft Versus Host Disease (cGVHD)
Brief Title: A Study of Belumosudil in Children With Chronic Graft Versus Host Disease (schoolROCK)
Acronym: schoolROCK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFI17893; U1111-1281-0103 (Registry Identifier: ICTRP); 2024-511508-18 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-07-25; First posted 2025-08-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- belumosudil (Experimental): Participant will take IMP with a meal approximately the same time each morning. IMP dose will be according to weight and will be increased to daily dose of twice a day (BID) in participants who concomitantly receive proton pump inhibitors (PPIs) or strong CYP3A4 inducers. No concomitant PPIs are allowed during Phase 1 up to and including Cycle 1 Day 15. From Day 16 onwards, PPIs will be permitted, resulting in an increased dose of Belumosudil to BID. No concomitant strong CYP3A4 inducers are allowed during Phase 1.
  Interventions: Drug: Belumosudil

INTERVENTIONS:
Drug: Belumosudil — Pharmaceutical form:Oral suspension -Route of administration:Oral or nasogastric tube
  Other Names: SAR445761; REZUROCK
Drug: Belumosudil — Pharmaceutical form:Tablet formulation-Route of administration:Oral
  Other Names: SAR445761; REZUROCK

SUMMARY:
This is an open-label, single group, Phase 1/2, 1-arm study for treatment of children aged 1 to <18 years with active moderate-to-severe cGVHD that is refractory to or recurred after at least 2 prior lines of systemic therapy for cGVHD.

The purpose of Phase 1 is to determine the PK profiles and to establish the Recommended Pediatric Equivalent Dose (RPED) of belumosudil in participants aged 1 to <12 years with active moderate to severe cGVHD. Upon completion and evaluation of Phase 1, Phase 2 will commence with the purpose of determining safety and efficacy (ORR by 24 weeks) of belumosudil in participants aged 1 to <18 years.

Study details include:

The end of study is defined as 3 years after the last participant is recruited or all participants have discontinued treatment, or have died, whichever comes first.

Minimum of 6 participants ages 1 to 6 years will be enrolled for each phase of study

Individual participant duration on study will consist of:

Up to 4 weeks for screening. Treatment until clinically significant progression of cGVHD, relapse/recurrence of the underlying disease, start of a new systemic treatment for cGVHD, experience of an unacceptable adverse event, request from participant or Investigator, or until the end of the study is reached, whichever comes first.

4 weeks of post treatment safety follow-up. Long-term follow-up until death or end of study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 1 to <18 years of age, at the time the consent/assent is signed. For Phase 1: participant must be 1 to <12 years of age, at the time the consent/assent is signed. For Phase 2: participant must be 1 to <18 years of age, at the time the consent/assent is signed.
* Participant has undergone an allogeneic HCT
* Has active moderate to severe cGVHD, defined using the NIH Consensus diagnosis and staging criteria for which systemic therapy is required
* cGVHD is refractory to or has recurred after at least 2 prior lines of systemic treatment
* Has received at least two lines of prior systemic therapy for cGVHD, but no more than 5 lines.
* If participant receives corticosteroid therapy for cGVHD, the dose must be stable for at least 2 weeks prior to the first dose of the IMP
* Has a Lansky-Play (if aged ≤16) or Karnofsky (if aged >16) performance scale of ≥60
* Body weight of 8 kg and above
* Contraceptive use by sexually active male and female should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Life expectancy of >6 months
* Participants can take the IMP orally or via a nasogastric tube

Exclusion Criteria:

* Progressive underlying disease or post-transplant lymphoproliferative disease within 4 weeks prior to the first dose of the IMP.
* Diagnosed with another malignancy (other than malignancy for which transplant was performed) within 3 years prior to the first dose of the IMP
* History or other evidence of severe illness or any other conditions that would make the participant, in the opinion of the Investigator, unsuitable for the study (such as malabsorption syndromes, active, uncontrolled infections, or poorly controlled psychiatric disease)
* Has a forced expiratory volume (in the first second; FEV1) ≤39% or has lung score of 3
* Female participants who are pregnant or breastfeeding
* Current treatment with systemic agents for cGVHD (apart from corticosteroids and calcineurin inhibitors), such as ibrutinib, ruxolitinib, sirolimus, mycophenolate (MMF), methotrexate, rituximab, imatinib, extracorporeal photopheresis (ECP) and any investigational cGVHD treatment. Prior treatment with these agents and/or therapy is allowed with a washout of at least 28 days or 5 half-lives, whichever is shorter, prior to the first dose of the IMP
* The use of herbal and recreational drugs within 7 days before the start of study intervention
* Participant has had previous exposure to belumosudil
* Administration of live or live-attenuated vaccines is prohibited within 28 days or 5 elimination half-lives of the respective vaccine, whichever is longer, prior to IMP administration and until study intervention discontinuation
* Treatment with any non-GVHD investigational agent, or any investigational device or procedure, within 28 days (or 5 half-lives, whichever is longer) of enrollment, prior to the first dose of the IMP
* For Phase 1 only: Administration with strong CYP3A4 inducers is not allowed within 14 days or 5 half-lives (whichever is longer) of the first dose of IMP until the study intervention discontinuation.
* For Phase 1 only: PPIs are not allowed within 1 day or 5 half-lives (whichever is longer) of the first dose of IMP and Day 15 of Cycle 1. They can be restarted on Cycle 1 Day 16.
* Absolute neutrophil count <1.0 × 109/L. The use of granulocyte-colony stimulating factor (G-CSF) is not allowed to reach this level during screening
* Platelet count <25 × 109/L. Platelet transfusions are not allowed within 72 hours before hematology screening test. Participants with platelet transfusion refractoriness will be excluded. (Participants who have suboptimal responses to at least 2 transfusions will be considered as platelet transfusion refractory)
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >3× upper limit of normal (ULN) (> 5x ULN if abnormalities are due to cGVHD)
* Total bilirubin >1.5 × ULN (>3 x ULN if Gilbert's syndrome)
* Glomerular filtration rate (GFR) <30 mL/min/1.73 m2 using the revised Bedside Schwartz calculator
* Participants with an active viral disease including hepatitis B virus (HBV) and hepatitis C virus (HCV)
* Active uncontrolled Cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infection
* Known history of human immunodeficiency virus (HIV)
* Not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2031-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Phase 1: AUC | Cycle 1 Day 15 after the last participant dosed in the phase 1 part.
  PK parameter (AUC at steady state)
Proportion of participants who achieve an overall response (partial response [PR] or complete response [CR]) by Week 25 or Cycle 7 Day 1 whichever is first | Up to 3 years after the last participant enrolled
  Proportion of participants who achieve an overall response (partial response [PR] or complete response [CR]) by Week 25 or Cycle 7 Day 1 whichever is first, as defined by the National Institute of Health (NIH) Consensus response criteria

SECONDARY OUTCOMES:
Phase 1: Number of participants with treatment-emergent adverse events [TEAEs], serious TEAEs, and adverse events of special interest (AESIs) | Up to 3 years after the last participant enrolled
  Safety
Phase 1: Cmax | Cycle 1 Day 15 after the last participant dosed in the phase 1 part
  Steady-state belumosudil PK parameters
Phase 1: AUC0-6h | Cycle 1 Day 15 after the last participant dosed in the phase 1 part
  Steady-state belumosudil PK parameters
Phase 1: ORR | Up to 3 years after the last participant enrolled
  Proportion of participants who achieve an overall response (complete response [CR] or partial response [PR]) by 24 weeks, as defined by the 2014 National Institute of Health (NIH) Consensus response criteria
Phase 1: DOR | Up to 3 years after the last participant enrolled
  Time from the date of first response to the date of progression of cGVHD, initiation of a new systemic treatment for cGVHD, or death, whichever comes first. DOR is determined only for participants who achieved overall response (PR or CR) as per 2014 NIH Consensus response criteria
Phase 1: response by organ | Up to 3 years after the last participant enrolled
  As defined by the 2014 NIH Consensus response criteria
Phase 1: failure-free survival (FFS) | Up to 3 years after the last participant enrolled
  Time from the date of the first investigational medicinal product (IMP) administration to the date of initiation of a new systemic treatment for cGVHD, relapse or recurrence of the underlying disease, or death, whichever occurs first
Phase 1: overall survival (OS) | Up to 3 years after the last participant enrolled
  Time from the date of first IMP administration to the date of death due to any cause
Phase 1: time to response (TTR) | Up to 3 years after the last participant enrolled
  Time from the date of the first IMP administration to the first documented response (either CR or PR) according to the 2014 NIH Consensus Criteria for cGVHD
Phase 2: Number of participants with treatment-emergent adverse events [TEAEs], serious TEAEs, and adverse events of special interest (AESIs) | Up to 3 years after the last participant enrolled
  Safety
Phase 2: Ctrough of belumosudil | Cycle 2 Day 1 and Cycle 4 Day 1 after the last participant enrolled
Phase 2: DOR | Up to 3 years after the last participant enrolled
  Time from first response to the date of progression of cGVHD, initiation of a new systemic treatment for cGVHD, or death, whichever comes first. DOR is determined only for participants who achieved overall response (PR or CR) as per NIH Consensus response criteria
Phase 2: response by organ | Up to 3 years after the last participant enrolled
  response by organ as defined by the 2014 NIH Consensus response criteria
Phase 2: FFS | Up to 3 years after the last participant enrolled
  Time from the date of the first IMP administration to the date of initiation of a new systemic treatment for cGVHD, relapse or recurrence of the underlying disease, or death, whichever occurs first
Phase 2: OS | Up to 3 years after the last participant enrolled
  Time from the date of first IMP administration to the date of death due to any cause
Phase 2: time to response (TTR) | Up to 3 years after the last participant enrolled
  Time from the date of the first IMP administration to the first documented response (either CR or PR) according to the 2014 NIH Consensus Criteria for cGVHD

CONTACTS AND LOCATIONS:
Locations (20):
- United States (2):
  - Memorial Sloan Kettering Cancer Center- Site Number : 8400001, New York, New York
  - Texas Children's Hospital - Baylor - PIN- Site Number : 8400008, Houston, Texas
- Belgium (2):
  - Investigational Site Number : 0560003, Ghent
  - Investigational Site Number : 0560001, Leuven
- China (3):
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560004, Shenzhen
  - Investigational Site Number : 1560002, Suzhou
- France (2):
  - Investigational Site Number : 2500002, Marseille
  - Investigational Site Number : 2500001, Paris
- Investigational Site Number : 2760001, Berlin, Germany
- Israel (4):
  - Investigational Site Number : 3760005, Haifa
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760001, Tel Aviv
  - Investigational Site Number : 3760003, Tel Litwinsky
- Investigational Site Number : 3800001, Roma, Italy
- Investigational Site Number : 5280001, Utrecht, Netherlands
- Spain (3):
  - Investigational Site Number : 7240003, Esplugues de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7240002, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240001, Barcelona
- Investigational Site Number : 8260002, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DFI17893 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26796&tenant=MT_SNY_9011